CLINICAL TRIAL: NCT00581022
Title: Assessment of Objective Sleep Disturbances in Orthostatic Intolerance
Brief Title: Objective Sleep Disturbances in Orthostatic Intolerance
Status: Completed | Type: Observational
Sponsor: Satish R. Raj (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Satish R. Raj, Assistant Professor of Medicine & Pharmacology, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 051131; UL1RR024975 (NIH)
Record Dates: First submitted 2007-12-22; First posted 2007-12-27 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Postural Tachycardia Syndrome; Chronic Orthostatic Intolerance
Keywords: postural tachycardia syndrome; sleep; insomnia
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with Chronic Orthostatic Intolerance
  Interventions: Procedure: Polysomnography

INTERVENTIONS:
Procedure: Polysomnography — Overnight Sleep Study
  Other Names: Sleep Study

SUMMARY:
We wish to study sleep architecture in patients with chronic orthostatic intolerance. We will test the null hypothesis that there is no difference in time during the various phases of sleep between patients and healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with chronic orthostatic intolerance (or healthy subject)

Exclusion Criteria:

* overt cause or acute orthostatic intolerance
* pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with chronic orthostatic intolerance by the Vanderbilt Autonomic Dysfunction Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Duration of sleep | 1 night

SECONDARY OUTCOMES:
Time in individual phases of sleep | 1 night
sleep latency | 1 might

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Unviersity, Nashville, Tennessee, United States